CLINICAL TRIAL: NCT00501332
Title: A Phase IIa, Open Label, Controlled, Dose Ranging Study of Maxy-G34 as an Adjunct to TAC Chemotherapy in High-Risk Patients With Stage I, II, or IIIa Breast Cancer.
Brief Title: Evaluation of Maxy-G34 in Breast Cancer Patients Treated With TAC (Docetaxel, Adriamycin, Cyclophosphamide) Chemotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maxygen Holdings Ltd. (Industry)
Collaborators: Maxygen ApS (Industry); Maxygen, Inc. (Industry); Parexel (Industry)
Responsible Party: Santosh Vetticaden, MD. Chief Medical Officer., Maxygen, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MP-CL-30166; EUDRACT No.: 2006-006565-16; PAREXEL 84728
Record Dates: First submitted 2007-07-12; First posted 2007-07-16 (Estimated); Last update posted 2007-12-24 (Estimated); Status verified 2007-12

CONDITIONS: Chemotherapy-Induced Neutropenia; Breast Cancer
Keywords: neutropenia; breast; cancer; chemotherapy
MeSH Terms: conditions — Breast Neoplasms; Neutropenia; Neoplasms | interventions — Maxy G34

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 2 (Active Comparator)
  Interventions: Biological: Maxy-G34

INTERVENTIONS:
Biological: Maxy-G34 — Maxy-G34 will be administered by subcutaneous injection during each of 6 TAC chemotherapy cycles.
  Other Names: pegylated recombinant human G-CSF

SUMMARY:
This is an investigation of the safety and efficacy of Maxy-G34 in breast cancer patients treated with TAC chemotherapy. Maxy-G34 will be given as a single injection during each cycle of chemotherapy, for a planned total of six chemotherapy cycles.

ELIGIBILITY:
Key Inclusion Criteria:

1. Males and females at least 18 years of age
2. Diagnosis of high-risk stage I, II or IIIa breast cancer suitable for adjuvant TAC chemotherapy as based on investigator judgment
3. Candidates for TAC chemotherapy, and no prior treatment with anthracyclines

Key Exclusion Criteria:

1. Received chemotherapy within last 3 month prior to screening, or expected to receive any chemotherapy other than TAC and / or immunotherapy between screening and 30 days after last planned study drug administration
2. Any clinically significant findings on history or examination that, in the opinion of the investigator, would preclude administration of TAC chemotherapy in the full dose, including abnormal liver function, inadequate cardiac function or clinically significant cardiac disease, neuropathy or other disease
3. Prior bone marrow or peripheral blood hematopoietic stem cell transplant
4. Any active cancer or history of prior malignancy within the last 5 years except carcinoma in situ of the cervix, basal cell carcinoma or squamous cell carcinoma of the skin or any surgically cured malignancy diagnosed 5 years or more before diagnosis of breast cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-07

PRIMARY OUTCOMES:
To determine the duration of grade 4 neutropenia after administration of Maxy-G34 in chemotherapy cycle 1. | over 1 cycle of TAC chemotherapy (approximately 3 weeks)

SECONDARY OUTCOMES:
To determine the duration of grade 4 neutropenia after administration of Maxy-G34 in chemotherapy cycles 2-6. | over cycles 2-6 of TAC chemotherapy (approximately from weeks 4-18)
To determine the incidence of grade 4 neutropenia after administration of each of the 6 doses of Maxy-G34. | over all 6 cycles of TAC chemotherapy (approximately 18 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Santosh Vetticaden, MD, Study Director — Maxygen, Inc.
Locations (15):
- Poland (3):
  - Bydgoszcz
  - Gdansk
  - Lublin
- Romania (5):
  - Alba Iulia
  - Bucharest
  - Jud. Bacau
  - Suceava
  - Timișoara
- Russia (5):
  - Leningrad Region
  - Moscow
  - Moscow Area
  - Ryazan
  - Saint Petersburg
- Ukraine (2):
  - Dnipropetrovsk
  - Uzhhorod